CLINICAL TRIAL: NCT05097014
Title: A Double Blind, Multicentre, Randomised, Placebo-Controlled, 3-Way Cross-Over Study To Evaluate The Effect Of A Triple Combination Of Beclometasone Dipropionate And Formoterol Fumarate Plus Glycopyrronium (CHF5993) And A Dual Combination Of Beclometasone Dipropionate Plus Formoterol Fumarate (CHF1535) Both Administered Via pMDI On Lung Hyperinflation And Exercise Endurance Time In Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: CHF5993 and CHF1535 pMDI on Lung Hyperinflation and Exercise Endurance Time in Subjects With COPD
Acronym: TRIFORCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-05993AA1-17; 2020-004718-36 (EudraCT Number)
Record Dates: First submitted 2021-10-12; First posted 2021-10-27 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung hyperinflation, exercise endurance time
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHF5993 (Active Comparator): pMDI fixed combination product of beclometasone dipropionate (BDP) 100 µg plus 6 µg of formoterol fumarate (FF) and 10 µg of glycopyrronium (G)
  Interventions: Drug: CHF5993
- CHF1535 (Active Comparator): pMDI fixed combination product beclometasone dipropionate (BDP) 100 µg plus 6 µg of formoterol fumarate (FF)
  Interventions: Drug: CHF1535
- Matched placebo (Placebo Comparator): Matched placebo pMDI
  Interventions: Other: Matched placebo

INTERVENTIONS:
Drug: CHF5993 — Pressurized metered dose inhaler (pMDI) 2 inhalations bid
  Other Names: TRIMBOW®
  Arms: CHF5993
Drug: CHF1535 — Pressurized metered dose inhaler (pMDI) 2 inhalations bid
  Other Names: FOSTER®
  Arms: CHF1535
Other: Matched placebo — Pressurized metered dose inhaler (pMDI) 2 inhalations bid
  Arms: Matched placebo

SUMMARY:
Double Blind, Multinational, Multicentre, Randomised, Placebo-Controlled, 3-Way Cross-Over Study To Evaluate The Effect Of A Triple Combination Of Beclometasone Dipropionate And Formoterol Fumarate Plus Glycopyrronium (CHF5993) And A Dual Combination Of Beclometasone Dipropionate Plus Formoterol Fumarate (CHF1535) Both Administered Via pMDI On Lung Hyperinflation And Exercise Endurance Time In Subjects With Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated written informed consent obtained prior to any study-related procedures.
2. Outpatient population.
3. Male or female subjects.
4. COPD diagnosis for at least 12 months before the Screening visit in accordance with the definition by the GOLD 2020 report.
5. Current or ex-smokers (who quit smoking for at least 6 months prior to Screening Visit) with a smoking history of at least 10 pack-years [pack-years = (number of cigarettes per day x number of years)/20]. E-cigarettes smoking cannot be used to calculate pack-year history.
6. A post-bronchodilator FEV1/FVC < 0.7 within 30 min after 4 puffs (4 x 100 µg) of salbutamol pMDI and a post-bronchodilator FEV1 ≥ 40% and <80% of the predicted normal values. If this is not met at screening, the test can be repeated once before randomisation.
7. Pre-bronchodilator functional residual capacity (FRC) of > 120% of predicted normal FRC values at Screening visit 1. If this criterion is not met at screening, the test can be repeated once before randomisation.
8. A score of >2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1.
9. Subjects on mono- or dual inhaled maintenance COPD treatment at a stable dose for at least 3 months prior to screening.
10. A cooperative attitude and ability to correctly use the study inhalers.
11. Female subjects must be women either of non-childbearing potential (WONCBP) defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile) or physiologically capable of becoming pregnant (i.e. women of childbearing potential (WOCBP)).

    Inclusion criteria assessed prior to Randomization:
12. CWRCE at Visit 1b: between 2 min and 11 min at 80% of maximum workload. In case the subject cycles for a shorter (i.e. < 2 min) or longer (i.e. > 11 min) period, the visit can be repeated with an adjusted workload once within a 1-week period.
13. Oxygen saturation (SpO2 measured by pulse oximeter) at least 82% during the incremental exercise test (IET) performed in the run-in period.
14. Subjects must be able to complete CWRCE at Visit 1b and then at Visit 2 without requirement for supplemental oxygen.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Known respiratory disorders other than COPD which may impact the efficacy of the study drug according the investigator's judgment. This can include but is not limited to current diagnosis of asthma, alfa-1 antitrypsin deficiency, active tuberculosis, lung cancer, severe bronchiectasis unrelated to COPD, sarcoidosis, lung fibrosis, pulmonary hypertension and interstitial lung disease.
3. Unstable concurrent disease: e.g. fever, uncontrolled hyperthyroidism, uncontrolled diabetes mellitus or other endocrine disease; significant hepatic impairment; significant renal impairment; uncontrolled gastrointestinal disease (e.g. active peptic ulcer); uncontrolled cardiac disease, uncontrolled neurological disease; uncontrolled haematological disease; uncontrolled autoimmune disorders, or other which may impact the efficacy or the safety of the study drug according to investigator's judgment.
4. Moderate (requiring prescriptions of systemic corticosteroids and/or antibiotics) or severe (leading to hospitalization) COPD exacerbation in the 3 and 12 months, respectively, prior to Screening visit 1 and during the run-in period.

8. Subjects requiring long term (> 15 hours a day) oxygen therapy for chronic hypoxemia.

5. Subjects who have clinically severe cardiovascular condition (such as but not limited to unstable ischemic heart disease, NYHA Class IV, left ventricular failure, myocardial infarction in the prior 6 months, not controlled arrhythmia etc.), which may impact the efficacy or the safety of the study drug according to the investigator's judgement.

6. An abnormal and clinically significant 12-lead electrocardiogram (ECG) which may impact the safety of the subject according to investigator's judgement. Subjects whose 12-lead ECG shows QTcF >450 ms for males or QTcF >470 ms for females at screening visit are not eligible.

7. History of hypersensitivity to M3 receptor antagonists, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the trial which may raise contra-indications or impact the efficacy of the study drug according to the investigator's judgement.

8. Subjects with serum potassium levels ≤ 3.5 mEq/L (or 3.5 mmol/L) 9. Subjects with body mass index less than 15 or greater than 35 kg/m2. 10. History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening visit.

11. Subjects with contraindications to cardiopulmonary exercise testing, including those whose exercise test is limited by non-respiratory or cardiovascular condition, e.g. by neurologic, orthopaedic, or other disorders.

12. Participation in another clinical trial where investigational drug was received less than 30 days or 5 half-lives whichever is longer prior to screening visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Inspiratory capacity (IC) prior to Constant Work Rate Cycle Ergometry (CWRCE) test | 3 weeks of treatment
  Change from baseline in 2-hour post-dose

SECONDARY OUTCOMES:
IC at Isotime, defined as the shortest CWRCE test duration among baseline and end of treatment period. | 3 weeks of treatment
  Change from baseline
Exercise endurance time (EET) | 3 weeks of treatment
  Change from baseline in 2-hour post-dose

OTHER OUTCOMES:
EET between CHF5993 and CHF1535 | 3 weeks of treatment
  Change from baseline in 2-hour post-dose
Pre-dose morning Forced Expiratory Volume in 1 second (FEV1) | 3 weeks of treatment
  Change from baseline
Pre-dose Forced Vital Capacity (FVC) | 3 weeks of treatment
  Change from baseline
Functional Residual Capacity (FRC) | 3 weeks of treatment
  Change from baseline in 2-hour post-dose
Pre-dose IC | 3 weeks of treatment
  Change from baseline
Residual Volume (RV) | 3 weeks of treatment
  Change from baseline in 2-hour post-dose
RV/Total Lung Capacitity (TLC) ratio | 3 weeks of treatment
  Change from baseline in 2-hour post-dose
Dyspnoea intensity at isotime (using the modified Borg scale) | 3 weeks of treatment
  Change from baseline
Physical activity (steps/day) | 3 weeks of treatment
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Watz, MD, Study Director — Pulmonary Research Institute at LungenClinic Grosshansdorf, German Center for Lung Research
Locations (1):
- PAREXEL International GmbH Early Phase Clinical Unit Berlin, Berlin-Spandau, Berlin Spandauer Damm, Germany

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Derived] Watz H, Kirsten AM, Ludwig-Sengpiel A, Krull M, Mroz RM, Georges G, Varoli G, Charretier R, Cortellini M, Vele A, Galkin D. Effects of inhaled beclometasone dipropionate/formoterol fumarate/glycopyrronium vs. beclometasone dipropionate/formoterol fumarate and placebo on lung hyperinflation and exercise endurance in chronic obstructive pulmonary disease: a randomised controlled trial. Respir Res. 2024 Oct 17;25(1):378. doi: 10.1186/s12931-024-02993-x. PMID 39420338